CLINICAL TRIAL: NCT01787656
Title: A Novel Method of Screening for Ovarian Cancer Using Gynecologic Fluids and Mucus
Status: Completed | Type: Observational
Sponsor: University of South Alabama (Other)
Collaborators: ProHealth Care, Inc (Other); Women's Cancer Care (Unknown); University of Tennessee Cancer Institute (Other); Arizona Oncology Associates (Network); Sarasota Memorial Hospital (Other); Florida Hospital Cancer Institute (Unknown); Crescent City Physicians, Inc. (Other); Sanford USD Medical Center (Unknown); Monongalia General Hospital (Unknown); Ochsner Health System (Other); Sacred Heart Health System (Other); Tennessee Valley Gynecologic Oncology (Unknown); Washington University School of Medicine (Other); Augusta University (Other); Tulane University Health Sciences Center (Other); Cancer Center of South Florida (Unknown); Mayo Clinic (Other); Marshall University (Other); Indiana University (Other); University of Arizona (Other); St. Luke's Hospital and Health Network, Pennsylvania (Other); Mercy Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: USA-MCI GON-1.01
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — De-idetified samples of gynecologic fluid, mucus, and blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Ovarian cancer is deadly and generally diagnosed at late stage when the chances of survival are low. There is a current belief that this cancer starts in the fallopian tubes and progresses towards the ovaries, spreading to the cells on the surface. Within the fallopian tubes and the uterus, there is a constant flow of mucus which has only one exit through the cervix and out the vagina. Proteins that are generated within the entire female reproductive system are trapped into this viscous fluid and eventually released as waste. When a routine PAP test is performed, a sample of this mucus is collected along with any cells, and preserved in the PAP fluid. The fluid is currently discarded but contains a protein profile showing of the status of the cells in the female reproductive system. We have examined this fluid and found that it contains unique peptides/proteins that provide a diagnosis of ovarian cancer when compared against healthy controls. These markers will be initially refined using the comparison of ovarian cancer patients against those with benign adnexal masses that entered the clinic during the same time period.

In this Phase II biomarker validation study we will further refine and validate these biomarkers using a new collection of samples from at least 200 ovarian cancer cases with epithelial ovarian cancer (endometroid and papillary serous histology, most common) and comparing these against 600 patients with a diagnosis of a benign adnexal mass that enter the clinics during the same time period. Patient samples will be collected on their first visit to the gynecologic oncologist at a number of collaborating clinics. Final processing of all of the samples will be performed within the proteomics research facilities of the Mitchell Cancer Institute using Selected Reaction Monitoring (SRM, with mass spectrometry) based on the refined set of makers statistically selected within the first aim. Biomarkers validated within this study will be compared with the well accepted CA-125 data for the patients. The research involves a three year validation and may allow detection of this cancer at a very early stage when the survival is as high as 90%. One aim examines a self-taken test that could allow its use in medically underrepresented and rural areas.

ELIGIBILITY:
Inclusion Criteria:

1. Must be fully consented to the collection of the samples in writing (completed consent forms).
2. Age Criteria: Women age 50 and older who are post menopausal (defined as 12 months past last menstrual period).
3. Must have: Diagnosis of an adnexal mass or a suspicion of ovarian cancer, or a suspected fallopian tube or primary peritoneal cancer.
4. Must have a uterus and cervix.
5. Surgery for the adnexal mass must be anticipated. (Only patients with an adnexal mass requiring surgery will be eligible).

Exclusion Criteria:

1. Any subject who has a condition that would increase the risk associated with the standard sampling procedures (Such as a pap smear, or cotton swab in vagina)
2. Prior hysterectomy.
3. Absence of adnexal mass.
4. Primary diagnosis of a cancer other than ovarian, primary peritoneal or fallopian tube.
5. Patients with grossly visible cervical cancer.
6. Previous/recent treatment for any invasive gynecologic cancer.
7. Recent chemotherapy within the prior 2 years. (recent neoadjuvant chemotherapy for ovarian cancer would exclude the patient from participation).
8. Cervical conization within the prior 6 months.
9. History of Radiation therapy to the pelvis, vagina or cervix.
10. Obvious advanced stage cancer (Stage III or IV) on presentation, if known prior to specimen collection.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with an adenxal mass or suspicion of ovarian, fallopian tube, or primary peritoneal cancer
Sampling Method: Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2013-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Discovery of biomarkers that allow for the early detection of ovarian cancer | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Finan, PhD, Principal Investigator — University of South Alabama
Locations (1):
- University of South Alabama Mitchell Cancer Institute, Mobile, Alabama, United States